CLINICAL TRIAL: NCT01336231
Title: Impact on Quality of Life, Fatigue and Cognitive Function in Anti-angiogenesis in Patients With Metastatic Kidney Cancer : a Pilot Study
Brief Title: Impact on Quality of Life, Fatigue and Cognitive Function in Anti-angiogenesis in Patients With Metastatic Kidney Cancer
Acronym: COG-ANGIO
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: COG-ANGIO
Record Dates: First submitted 2011-04-12; First posted 2011-04-15 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Kidney Cancer
Keywords: quality of life; cognitive functions; antiangiogenic agents; kidney cancer; metastatic
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients group: Patients with a metastatic kidney cancer and must beginning a treatment by antiangiogenic

SUMMARY:
Longitudinal study nonrandomized, multicenter observational descriptive monitoring patients treated with anti-angiogenic for metastatic kidney cancer

ELIGIBILITY:
Inclusion Criteria:

* Patient (e) Age (e) over 18 years
* Kidney cancer metastatic or locally advanced
* Anti-angiogenic or targeted therapy (bevacizumab, sorafenib, sunitinib, temsirolimus, another molecule or developing or having obtained authorization in this indication) may be associated with interferon or combined together
* Proposed treatment in first line or second line
* Brain imaging not finding brain metastases
* Having signed the informed consent of study participation
* The patient may have received prior anti-angiogenic

Exclusion Criteria:

* Cancer of the kidney other than primitive
* Previous history of cancer other than kidney cancer in complete remission for less than 5 years
* Patients under 18 years
* Patients whose treatment is associated with chemotherapy
* disorders of cognitive functions to existing treatment delivery
* Pathology psychiatric evolutionary
* Refusal of participation
* Patient unable to respond to cognitive tests
* Drug use
* Heavy drinking (WHO criteria)
* History of stroke
* History of head trauma
* Brain metastases known
* MMS below normal compared to existing standards for age and socio-cultural

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a metastatic kidney cancer and must beginning a treatment by antiangiogenic
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2008-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Impact of fatigue, memory problems and attentional | up to 12 months after treatment
  Assessing the impact of fatigue, memory problems and attentional induced by an anti-angiogenic and study their evolution over time in patients with metastatic kidney cancer.

SECONDARY OUTCOMES:
Parameters of quality of life | up to 12 months after treatment
  Studying the different parameters of quality of life and their evolution over time.
disorders of cognitive functions | up to 12 months after treatment
  Studying the correlations between disorders of cognitive functions and parameters of quality of life and fatigue.
biological disturbances | up to 9 months after treatment
  Search for biological disturbances may be related to fatigue and cognitive disorders.
Impact of anxiety and depression | up to 12 months after treatment
  Assessing the impact of anxiety and depression at the waning of treatment
List of symptoms | up to 12 months after treatment
  Compare the list of symptoms considered important by the patient compared to those recorded in the medical record.
Impact on the sexuality | up to 12 months after treatment
  sess the impact on the sexuality of patients with the waning of treatment
Effects of different antiangiogenic agents | up to 12 months after treatment
  Compare the impact on quality of life and cognition side effects of different antiangiogenic agents used

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY-LOBBEDEZ, PD, Principal Investigator — Centre François Baclesse
Locations (6):
- France (6):
  - Centre François BACLESSE, Caen, Calvados
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - CHU, Rouen, Seine Maritime
  - CHU, Strasbourg
  - Institut Gustave Roussy, Villejuif
  - Hôpital Georges Pompidou, Paris, Île-de-France Region